CLINICAL TRIAL: NCT06950632
Title: Effect of Peppermint Oil Inhalation on Intensity and Frequency of Acute Nausea and Vomiting in Cancer Patients Receiving Chemotherapy: A Randomized Controlled Trial
Brief Title: This Study Will Investigate the Effectiveness of Peppermint Oil Inhalation in Reducing the Intensity and Frequency of Acute Nausea and Vomiting Among Cancer Patients Undergoing Chemotherapy. Chemotherapy-induced Nausea and Vomiting (CINV) Are Among the Most Distressing Side Effects Experienced by pa
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, QURAT-UL-AIN, Qurat-Ul-Ain, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Institute of Nursing
Record Dates: First submitted 2025-04-22; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Chemotherapy Induced Nausea and Vomiting
Keywords: Peppermint oil inhalation
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peppermint oil inhalation (Experimental): Participants in the experimental group will inhale five drops of 100% pure peppermint essential oil placed on a cotton ball inside a container for ten minutes before each chemotherapy session and every two hours during the infusion
  Interventions: Dietary Supplement: Pepppermint oil inhalation
- Control group (Sham Comparator): The control group will inhale five drops of distilled water placed on a cotton ball inside a container for ten minutes before each chemotherapy session and every two hours during the infusion
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Pepppermint oil inhalation — Participants in the experimental group will inhale five drops of 100% pure peppermint essential oil placed on a cotton ball inside a container for ten minutes before each chemotherapy session and every two hours during the chemotherapy infusion.
  Arms: Peppermint oil inhalation
Dietary Supplement: Placebo — The control group will follow the same procedure using five drops of distilled water placed on a cotton ball inside a container for ten minutes before each chemotherapy session and every two hours during the infusion
  Arms: Control group

SUMMARY:
Cancer is a major cause of death and disability worldwide and in South Asian countries. Cancer treatment options include chemotherapy, radiation therapy, surgery, and adjuvant therapy (Additional treatments after primary cancer treatment such as surgery, radiation, or chemotherapy are used to lower the chance of cancer recurrence or remove any remaining cancer cells). Chemotherapy poses serious adverse effects, including fatigue, hair loss, skin irritation, loss of appetite, change in bowel habits, weakened immune system, dry mouth, peripheral neuropathy, nausea and vomiting. Chemotherapy-induced nausea and vomiting cause fluid-electrolyte imbalance, dehydration, weight loss and physiological consequences due to inadequate medication absorption or compromised kidney clearance. Although anti-emetic drugs are given to reduce CINV but these drugs pose some serious adverse effects including heartburn, insomnia, headache, dizziness, constipation/diarrhea, loss of muscle control, pharyngeal itching, dry mouth and also increases economic burden on the patient and his/her family. The limited and hazardous side effects of these medications have led to a shift towards non-pharmacological and home remedies. Using natural remedies is a simple and low-risk measure in this regard. This study aims to evaluate the effects of peppermint oil inhalation on the intensity and frequency of Chemotherapy induced acute nausea and vomiting among cancer patients undergoing chemotherapy. A randomized controlled trial will be conducted using non-probability convenience sampling, followed by random assignment to intervention and control groups. The target population comprises patients receiving chemotherapy at the outpatient oncology department of Jinnah Hospital, Lahore. A total of 106 patients will be enrolled. The intervention group will receive peppermint oil inhalation, while the control group will receive a placebo. Descriptive statistics (frequency, percentage, mean, and standard deviation) will be used to summarize participant's characteristics. Chi-square test will be applied to compare demographic variables (e.g., age, gender, marital status, education, occupation, and RINV categories) between groups. An independent t-test will be used to compare the mean RINV scores post-intervention between intervention and control group. A p-value of <0.05 will be considered statistically significant. It is anticipated that peppermint oil inhalation will significantly reduce the severity and frequency of Chemotherapy induced acute nausea and vomiting. If effective, this complementary intervention could offer a low-cost, safe alternative to supplement standard anti-emetic therapies, potentially easing the financial and physiological burden associated with pharmacological treatments.

ELIGIBILITY:
Inclusion Criteria:

* • Participants undergoing chemotherapy in the outpatient oncology department of Jinnah Hospital Lahore.

  * Participants ages 20-50 years.
  * Participants of Both genders' male and female.
  * Participants who have undergone under one cycle of chemotherapy.
  * Participants who can understand and comprehend Urdu and Punjabi language

Exclusion Criteria:

* Participants who are allergic to peppermint products.
* Participants who have any psychiatric illness.
* Participants diagnosed with any respiratory illness.
* Participants who have vomiting due to any ailment other than chemotherapy.
* Participants with Gastro-intestinal and Hepatobiliary Tumors.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-10-20 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Effect of Peppermint Oil Inhalation on the Intensity and Frequency of Acute Nausea and Vomiting Measured by RINV Scale | Within 24 hours after chemotherapy (acute phase)
  The primary outcome is the change in the intensity and frequency of acute nausea and vomiting, assessed by the Rhodes Index of Nausea, Vomiting, and Retching (RINV) Scale, within 24 hours following chemotherapy. Comparison of mean RINV scores will be made between the experimental (peppermint oil inhalation) group and the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Jinnah Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided